CLINICAL TRIAL: NCT03719976
Title: Prepared Parents Helping Kids: Teaching Health Care Navigation for Bhutanese Parents
Brief Title: Prepared Parents Helping Kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-015474; 1K23HD082312-01A1 (NIH)
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Immigrant Caregiver Health Care Navigation for Children
Keywords: Refugee Health; Immigrant Health; Health care navigation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthcare navigation workshops (Experimental): All enrolled caregivers and parents will partake in the group-based educational intervention.
  Interventions: Other: Group-based educational intervention

INTERVENTIONS:
Other: Group-based educational intervention — The group-based educational intervention will use a bilingual Community Health Worker (CHW) who will teach parents key skills needed to access health care for children. Parents will be invited to attend 6 small, closed-group sessions held over 12 weeks and lasting no more than 75 minutes. Sessions will be interactive, culturally-appropriate, and held in parents' preferred language.

SUMMARY:
Learning to navigate the US health system is challenging for many new immigrants. This pilot study will determine whether an intervention to teach parents key skills needed to access health care for children is feasible and acceptable to immigrant parents.

This study will also look for evidence of efficacy to inform the planning process for future, larger evaluations of the intervention (i.e., estimate effect sizes).

DETAILED DESCRIPTION:
Parents-particularly those with limited English proficiency (LEP) and limited literacy-may require months or years of experiential learning to master fundamental health care navigation tasks, such as requesting an interpreter. Most programs teaching health care navigation skills are ad hoc and have not be evaluated.

In this study, Investigators will pilot a group-based educational intervention in which a bilingual community health worker will use an interactive curriculum to teach immigrant parents key skills needed to access health care for children.

Parents and caregivers for children <18 years will be enrolled in closed groups of 6-12 individuals. The 6-12 week intervention will comprise 6 meetings, each of which will be no longer than 75 minutes. Each meeting will focus on one of six skills:

1. Requesting an interpreter;
2. Communicating with a health care facility by telephone;
3. Scheduling appointments;
4. Traveling to health care facilities and registering with the front desk;
5. Obtaining appointments with specialists;
6. Calling 911 for an ambulance.

Each meeting will follow a pre-specified plan that will typically include welcoming activities, a review of prior material, introduction of new material, and a series of activities (e.g., role play) to practice key skills. Sessions will be interactive, culturally-appropriate, and held in parents' preferred language.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 years or older
* Parent of a child <18 years
* Nepali-speaking
* Resident of the US for <10 years

Exclusion Criteria:

* Scheduled to move away from the study location (e.g., to another city) before the end of the 6-session intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects enrolling in study and completing study visits | 9 months
  Enrollment of the target sample and completion of the planned study visits by participants

SECONDARY OUTCOMES:
Change in retainment of health care navigation skills from baseline | 9 months
  Change in Health Care Navigation Inventory (HCNI) Skills Subscale scores from baseline to post-intervention study visits. Scores can range from 12 to 60, with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Yun, MD MHS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Bhutanese American Organization - Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No